CLINICAL TRIAL: NCT05394441
Title: Selected Health and Quality of Life Indicators Among ITMO University Students, Faculty and Staff
Brief Title: Health and Quality of Life of ITMO University's Students, Faculty and Staff
Status: Completed | Type: Observational
Sponsor: ITMO University (Other)
Responsible Party: Sponsor
Other Study IDs: 922022/4.3.1
Record Dates: First submitted 2022-05-24; First posted 2022-05-27 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Quality of Life
Keywords: students; faculty; academia; university

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — plasma samples will be collected and saved
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy adults (16+): Healthy students, faculty and staff of ITMO University older than 16 years

SUMMARY:
This study assess various indicators of physical and mental health, quality of life, well-being and satisfaction among students, faculty and staff of ITMO University. Participants are invited to join the study via informational web-site. Several quality of life indicators are obtained via surveys and some blood samples are taken to assess health condition.

DETAILED DESCRIPTION:
Students, faculty and staff from ITMO University are invited to participate in health examination on the campus. Surveys, such as EQ-5D-5L, K10+OHQ29, PSQI and others, assess different aspects of quality of life related to health. Also participants are asked to undergo several measurements by the interviewer (waist, hips, height, weight and others). Moreover blood samples are taken from the participants and lipidogram, cholesterol and glycohemoglobin are checked.

ELIGIBILITY:
Inclusion Criteria:

* student, faculty or staff from ITMO University
* participants, who signed informed consent and consent for data gathering
* participants, who signed consent to enroll in following surveys and health check-ups

Exclusion Criteria:

* participants younger than 16 years old
* participants with acute conditions distorting quality of life assessment
* participants, who did not sign informed consent and consent for data gathering - participants, who did not sign consent to enroll in following surveys and health check-ups

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Students, faculty and staff from ITMO University
Sampling Method: Non-Probability Sample
Enrollment: 830 (Actual)
Dates: Start 2022-06-02 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Cholesterol | 30 days
  Measured by A15 biochemical automatic analyzer (Biosystem, Spain)
Lipidogram | 30 days
  Measured by A15 biochemical automatic analyzer (Biosystem, Spain)
Glycohemoglobin | 30 days
  Measured by Architect c8000
Distress | 30 days
  Global measure of distress based on questions about anxiety and depressive symptoms that a person has experienced in the most recent 4 week period measured by Kessler-10 questionnaire
Psychological well-being | 30 days
  Measured by Oxford Happiness Questionnaire (OHQ)
Health status and quality of life | 30 days
  Measured by EuroQOL-5 Dimension Questionnaire (EQ-5D-5L)
Nicotine dependence | 30 days
  Nicotine dependence across all nicotine product types including cigarettes and electronic cigarettes measured by The Penn State Nicotine Dependence Index
Diabetes risk score | 30 days
  The 10-year risk of type 2 diabetes mellitus (DM), including asymptomatic diabetes mellitus and impaired glucose tolerance (IGT) measured by The Finnish Diabetes Risk Score
Sleep quality and disturbances. | 30 days
  Measured by Pittsburgh Sleep Quality Index
Physical activity | 30 days
  The types of intensity of physical activity and sitting time that people do as part of their daily lives measured by International Physical Activity Questionnaire - Short Form
Emotional eating, external eating, and restrained eating behavior | 30 days
  Qualitative and quantitative assessment of eating disorders associated with overeating and accompanying obesity measured by Dutch Eating Behavior Questionnaire
Alcohol use | 30 days
  Problematic alcohol use, including possible alcohol use disorders measured by The Russian version of the Alcohol Use Disorders Identification Test (AUDIT)
Ischemic heart disease prediction | 30 days
  Measured by The Rose angina screening questionnaire
Retinopathy | 30 days
  Measured with non-mydriatic fundus camera
Ocular fundus condition | 30 days
  Measured with non-mydriatic fundus camera

CONTACTS AND LOCATIONS:
Locations (1):
- ITMO University, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: Undecided